CLINICAL TRIAL: NCT01633190
Title: Canadian Rotavirus Surveillance Through the Immunization Monitoring Program Active (IMPACT): Assessment of Hospitalizations and Emergency Department Visits - the Impact of Publicly Funded Vaccine Programs in Canada
Brief Title: Canadian Rotavirus Surveillance Through the Immunization Monitoring Program Active (IMPACT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Canadian Paediatric Society (Other)
Responsible Party: Sponsor
Other Study IDs: ROTA 2010-2017
Record Dates: First submitted 2012-06-12; First posted 2012-07-04 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Viral Gastroenteritis Due to Rotavirus
Keywords: Surveillance; Rotavirus; Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rotavirus: - Children (0-16 years of age)admitted to hospital (through to December 31, 2020)

SUMMARY:
* Rotavirus Hospital Admissions Surveillance
* Retrospective surveillance for 2010 and 2011 for hospital admissions in children aged 0 to 16 years due to rotavirus gastroenteritis will be completed by all centers of the IMPACT (Immunization Monitoring Program, ACTive) pediatric hospital network.
* Prospective surveillance of rotavirus-related admissions for children aged 0 to 16 years was conducted in 2012-20 inclusive and will be performed for an additional 2 years until the end of 2022 at all 12 sites. Surveillance methodology will continue using the same case-finding strategy and the same case report form as in past surveillance (Case reporting is done electronically.
* Emergency Department Burden of Disease Case finding for all-cause diarrheal illness using ICD codes was undertaken prospectively for 2012 to 2014 and will not continue in the years 2015-17 inclusive. Systematic stool sampling was carried out for cases of gastroenteritis in children < 5 years of age presenting to the ED departments at the IMPACT hospitals in 2012 and 2013 and 5 of the 12 center hospitals in 2014. This component will not continue in to the 2015-17 protocol study years. However the admitted cases presenting to the IMPACT center hospitals with positive rotavirus will be reported and stool samples saved for genotyping at a later date.

DETAILED DESCRIPTION:
This study has the ability to provide contemporary Canadian data on the two of the most important outcome measures for effectiveness of rotavirus vaccine: hospital admissions and emergency department visits. The extended time period that already exists prior to vaccine implementation (2005 to 2017) will provide longterm baseline data with which to compare disease burden from 2012 to 2022.

The major advantages to this study are that surveillance occurs at the same hospitals and the same methodology and CRF has been used since 2005. This will ensure reliability and consistency in the surveillance study. The national data set captures patients from age group 0 to 16 years in 12 centers across the country. The retrospective and prospective studies will be in a unique position to capture all children admitted to the 12 pediatric hospitals in Canada. Since reliance on discharge codes alone may underestimate gastroenteritis due to rotavirus, laboratory surveillance coupled with medical record review will ensure the complete capture of the true disease burden. Data on the health status of children will facilitate the evaluation of children who are medically fragile for which rotavirus infections may be more significant.

ELIGIBILITY:
There are two parts to this criteria- Hospital admission surveillance (to December 31, 2019); and genotype surveillance (to December 31, 2020)

Hospital admission surveillance:

Inclusion Criteria:

* Age 0 to 16 years of age.
* Inpatient status at the IMPACT hospital
* Acute onset of symptoms of acute gastroenteritis with or without diarrheal stools, with or without vomiting, with or without fever.
* Laboratory confirmation of rotavirus in stool specimens or autopsy tissue sample with the use of antigen detection methods (enzyme linked immunoassay [ELISA] or immunochromatographic methods) or electron microscopy or molecular (PCR) diagnosis in a stool specimen taken within 14 days after the onset of gastrointestinal symptoms. Cases identified by autopsy must have had gastrointestinal symptoms before death.
* Referred cases of rotavirus infections that have laboratory confirmation from another institution using the same criteria as above

Exclusion criteria

* Non-laboratory confirmed diagnosis.
* Clinical data is not accessible to the nurse monitor.
* Incidental findings of rotavirus in patients admitted to hospital without acute gastrointestinal symptoms.

Rotavirus Genotype Surveillance - on stool sample already obtained for hospital admission purposes (not additional for the surveillance).

- Rotavirus identification: Rotavirus identification at sites will be accomplished by rotavirus antigen detected by EIA (Enzyme Immuno Assay) or electron microscopy.

Ages: 1 Minute to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children age 0-16 admitted to the participating IMPACT hospitals (to December 31, 2020) with confirmation of positive stool samples.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2012-03; Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
- Changes in rotavirus hospitalization rates in 12 pediatric hospitals in Canada pre- and post rotavirus vaccine implementation within publicly funded provincial programs | Patients are identified on admission starting January 1, 2018. The surveillance period begins when rotavirus is identified and continues until the patients are discharged (average 3-4 days). The study end date is December 31, 2020
  Described In the title

SECONDARY OUTCOMES:
- The number of hospital acquired rotavirus infections in children compared pre- and post immunization burden across the network. | Patients are enrolled when rotavirus is identified on a hospitalized patient. The patient is followed until discharge or symptoms of infection have ceased (average 5 days). Enrolment starts January 1, 2012 and ends December 31, 2020.
  Described in the title
- The most common rotavirus genotypes in hospitalized patients | Stool specimens from 2012 to 2020 will be collected at the time of laboratory diagnosis. Collection of isolates starts January 1, 2012 and continues to December 2020.
  Described in the title

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Le Saux, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (12):
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Winnipeg Children's Hospital, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Center, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU Sainte-Justine Hospital, Montreal, Quebec
  - Centre Mère-Enfant de Québec -Pavillon CHUL, Ste Foy, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IMPACT general web site — http://www.cps.ca/en/impact